CLINICAL TRIAL: NCT03678350
Title: Light Dosimetry for Intraoperative Photodynamic Therapy (IO-PDT) With Porfimer Sodium (Photofrin) in Patients With Malignant Mesothelioma or Non-Small Cell Lung Cancer (NSCLC), or Other Malignancies With Pleural Disease - Phase I Study
Brief Title: Light Dosimetry for Photodynamic Therapy With Porfimer Sodium in Treating Participants With Malignant Mesothelioma or Non-Small Cell Lung Cancer With Pleural Disease Undergoing Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Lumeda,Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 62118; NCI-2018-01663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 62118 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-08-30; First posted 2018-09-19 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Malignant Mesothelioma; Non-Small Cell Lung Carcinoma; Pleural Disorder
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Pleural Diseases | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Dihematoporphyrin Ether; Trioxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (porfimer sodium, IO-PDT) (Experimental): Participants receive porfimer sodium IV over 3-5 minutes and receive IO-PDT via a light dosimetry system 24-48 hours later.
  Interventions: Device: Light Dosimetry for Intranoperative Therapy; Procedure: Photodynamic Therapy; Drug: Porfimer Sodium

INTERVENTIONS:
Device: Light Dosimetry for Intranoperative Therapy — Undergo IO-PDT
Procedure: Photodynamic Therapy — Undergo IO-PDT
  Other Names: PDT; Photoradiation Therapy
Drug: Porfimer Sodium — Given IV
  Other Names: CL-184116; DHE; Dihematoporphyrin Ester; dihematoporphyrin ether; Photofrin II

SUMMARY:
This phase I trial studies the side effects and how well light dosimetry system works during photodynamic therapy with porfimer sodium in treating participants with malignant mesothelioma , non-small cell lung cancer or any other malignancy with pleural disease undergoing surgery. Light dosimetry measures the amount of laser light given during photodynamic therapy. Photodynamic therapy uses a drug, such as porfimer sodium, that becomes active when it is exposed to light. The activated drug may kill tumor cells. Using light dosimetry for intraoperative photodynamic therapy may help doctors estimate how much light is delivered during photodynamic therapy and decide if the treatment should be stopped or continued.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that our light dosimetry system is safe and effective in guiding intraoperative photodynamic therapy with porfimer sodium (Photofrin).

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (PFS) and overall survival (OS). II. To examine the relationship between immune biomarkers and response.

OUTLINE:

Participants receive porfimer sodium intravenously (IV) over 3-5 minutes and receive intraoperative photodynamic therapy (IO-PDT) via a light dosimetry system 24-48 hours later.

After conclusion of study treatment, participants are followed up at 30 days, within 4 weeks from surgery and PDT and every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant mesothelioma , non-small cell lung cancer (NSCLC) or other malignancies with pleural disease without distant disease.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) scale of 0-2.
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months after surgery. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* The subject must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent prior to receiving any study related procedure.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* White blood cell (WBC) < 4,000.
* Platelet count < 100,000.
* Total serum bilirubin > 2 mg/dL.
* Serum creatinine > 2 mg/dL.
* Alkaline phosphatase > 3 times the upper normal limit.
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 3 times the upper normal limit.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female subjects.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator?s opinion deems the subject an unsuitable candidate to receive porfimer sodium.
* Received an investigational agent within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 | Up to 30 days
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles. All subjects who receive any study treatment will be considered evaluable for toxicity.

SECONDARY OUTCOMES:
Progression-free survival | From time of surgery + photodynamic therapy (PDT) or, until start of a new treatment, disease progression or death (whichever occurs first), assessed up to 3 years
  The estimated distribution of progression free survival will be obtained using the Kaplan-Meier method. Estimates of quantities such as median survival will be obtained. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Overall survival (OS) | From the time of treatment (surgery + PDT) until death from any cause, assessed up to 3 years
  Estimates of quantities such as median survival will be obtained. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Anti tumor response | Up to 2 years
  Monitor immune markers for correlation between the IO PDT treatments and local or distant disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Saikrishna Yendamuri, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States